CLINICAL TRIAL: NCT03882788
Title: Anesthesia and the Developing Brain: a Comparison of Two Anesthetic Techniques
Brief Title: The Effect of Anesthesia on Neurodevelopmental Outcome (NDO)
Acronym: NDO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: The Gerber Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: NDO
Record Dates: First submitted 2016-05-05; First posted 2019-03-20 (Actual); Results first posted 2022-05-09 (Actual); Last update posted 2022-05-09 (Actual); Status verified 2022-05

CONDITIONS: Anesthesia; Adverse Effect; Congenital Heart Disease; Neurodevelopmental Disorders
MeSH Terms: conditions — Heart Defects, Congenital; Neurodevelopmental Disorders | interventions — Isoflurane; Fentanyl

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: EEG, metabolic/NMRS analysis and neurodevelopment outcome is blinded.
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Volatile Anesthesia (Active Comparator): In volatile anesthetic technique, maintenance of anesthesia will be standardized to the anesthesia will be standardized to the volatile anesthetic isoflurane.
  Rocuronium or pancuronium will be used for muscle relaxation. Additionally, narcotic fentanyl will be administered at no greater than 2 mcg/kg/hr (low dose). However, the primary anesthetic during CPB will be isoflurane with no narcotic administered during CPB.
  Interventions: Drug: Isoflurane; Drug: Fentanyl (low dose)
- Narcotic based anesthesia (Active Comparator): In narcotic based anesthetic technique, no volatile anesthetics will be used past induction.
  Maintenance of anesthesia will be with fentanyl 5 mcg/kg/hr not to exceed 10 mcg/kg/hr (high dose).
  Interventions: Drug: Fentanyl (high dose)

INTERVENTIONS:
Drug: Isoflurane — Isoflurane (volatile anesthesia) will be delivered at 1.5-2.0%% as required for anesthetic management.
  Arms: Volatile Anesthesia
Drug: Fentanyl (high dose) — Fentanyl (narcotic anesthesia) maintenance will be with fentanyl 5 mcg/kg/hr not to exceed 10 mcg/kg/hr.
  Arms: Narcotic based anesthesia
Drug: Fentanyl (low dose) — Fentanyl (narcotic anesthesia) maintenance will be with fentanyl 2 mcg/kg/hr.
  Arms: Volatile Anesthesia

SUMMARY:
The purpose of this study is to assess whether the type of anesthesia, narcotic-based versus inhalational anesthesia administered during cardiopulmonary bypass (CPB) surgery contributes to the wide variation in neurologic recovery and developmental outcome after surgery in infants with congenital heart disease.

DETAILED DESCRIPTION:
All subjects will be consented prior to participation in this study and prior to randomization.

All the subjects enrolled in the study will receive a preoperative assessment by one of the cardiac anesthesiologists and receive standardized induction with sevoflurane up to 2%, 2 mcg/kg of fentanyl and 1 mg/kg of rocuronium. The anesthetic maintenance will be determined using a computer- generated randomization table and assigning each patient to one of the two anesthetic regimens. Both of these anesthetic techniques are standard of care and are commonly used for these procedures.

Anesthetic Technique:

Volatile anesthetic:

In volatile anesthetic technique, maintenance of anesthesia will be standardized to the volatile anesthetic isoflurane. Isoflurane will be used for the study since this is what is presently available on the CPB machines. Anesthesia at 1.0 minimum anesthetic concentration (MAC) indicates that at this concentration 50% of the patients will not move when surgically stimulated. Anesthesiologists commonly use about 1.2-1.4 MAC in neonates, since the MAC value in infants is higher than that of children and adults. Isoflurane will be delivered at 1.5-2.0%% as required for anesthetic management.

Rocuronium or pancuronium will be used for muscle relaxation. Narcotic, fentanyl will be administered at no greater than 2 mcg/kg/hr.

Narcotic-based anesthetic:

In narcotic based anesthetic technique, no volatile anesthetics will be used except during induction.

Maintenance of anesthesia will be with fentanyl 5 mcg/kg/hr not to exceed 10 mcg/kg/hr.

The anesthetic may be supplemented with dexmedetomidine 0.05 mcg/kg/hr but not to exceed 1.0 mcg/kg/hr. Narcotic-based anesthetic will be used by the cardiac anesthesia team and the CPB technician throughout the operative case. 5 mcg/kg/hr of fentanyl is felt to represent 0.6 MAC of anesthesia.

Postoperative Sedative and Analgesic Care:

As per institutional standard of care, postoperative sedation will consist of fentanyl infusions of 2-4 mcg/kg/hr for the first 48 hours postoperatively.

A total of 9 Blood samples will be collected at different time points throughout the entire study for metabolomics determination (NAA/Cr and Chol/Cr)

EEG monitoring will be done for baseline in the pre-operative period for 15-20 minutes, during surgery and post-operatively up to 48 hours and prior to discharge for 15-20 minutes. Neurological and behavioral testing including Bayley Exam III will be done at 18-48 months.

ELIGIBILITY:
Inclusion Criteria:

* Neonates of at least 32 weeks of gestation, infants and children up to 2 years of age admitted to The Children's Hospital for treatment of cyanotic or non-cyanotic heart disease requiring surgical intervention.
* Admitting diagnosis of cyanotic or non-cyanotic heart disease

Exclusion Criteria:

* Neonates less than 32 weeks of gestational age, and children more than 2 years of age.
* Any documented central nervous system malformations.
* Any potential subject requiring unexpected postoperative Extracorporeal membrane oxygenation (ECMO) support

Ages: 1 Day to 36 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 153 (Actual)
Dates: Start 2013-04-22 (Actual); Primary Completion 2020-11-19 (Actual); Study Completion 2020-11-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lisa W Faberowski, MD, MSc, Principal Investigator — Stanford University
Locations (1):
- Stanford Childrens hospital, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: No
No IPD will be shared with other researchers

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Randomization data are available for only 89 of the 153 participants enrolled.
Groups:
- Narcotic Based Anesthesia: Participants receive fentanyl 5 mcg/kg/hr not to exceed 10 mcg/kg/hr (high dose).
- Volatile Anesthesia: Participants receive volatile anesthetic isoflurane (1.5-2.0%) as primary anesthetic; participants also receive rocuronium or pancuronium for muscle relaxation, and fentanyl at no greater than 2 mcg/kg/hr (low dose).
Period: Overall Study
Arm/Group | Narcotic Based Anesthesia | Volatile Anesthesia
Started | 44 | 45
Completed | 44 | 45
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Participants with randomization data are included in the analysis.
Groups:
- Total: Total of all reporting groups
Arm/Group | Narcotic Based Anesthesia | Volatile Anesthesia | Total
Number analyzed (Participants) | 44 | 45 | 89
Age, Continuous [Mean (Standard Deviation); unit: months] | 8.1 (8.5) | 6.2 (8.5) | 7.1 (8.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 20 | 38
  Male | 26 | 25 | 51
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 20 | 18 | 38
  Black or African American | 1 | 2 | 3
  Asian | 9 | 8 | 17
  Hispanic | 14 | 15 | 29
  Native Hawaiian or Other Pacific Highlander | 0 | 2 | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 44 | 45 | 89

OUTCOME MEASURES:

1. Primary Outcome: Bayley III
Description: Neurodevelopmental assessment scores are age dependent and based motor and behavioral abilities, often reported for normal or abnormal for age. Bayley Scales of Infant and Toddler Development, third edition, (Bayley III) is an instrument designed to measure the developmental functioning of infants and toddlers between the ages of 1 month and 42 months (age adjustments for prematurity are accommodated with the tool). It provides age specific composite scores for cognitive (91 items, score min 55 max 145), language (98 items, score min 47 max 153), and motor (138 items, score min 46 max 154) skills. For all scales, higher scores are better and lower scores indicate possible delay/deficit.
Time Frame: Assessed once between age 18 to 48 months (approximately 2 hours to assess), up to 48 months from study start
Population: Participants with a completed Bayley III assessment are included in the analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Narcotic Based Anesthesia | Volatile Anesthesia
Number analyzed (Participants) | 10 | 18
score on a scale
  Cognitive Standard Score | 91 (10) | 93 (15)
  Language Standard Score | 88 (11) | 90 (18)
  Motor Standard Score | 97 (13) | 90 (15)

2. Primary Outcome: Electroencephalogram
Description: Brain electrical activity: observation is for brain region specific abnormal or seizure activity. Number of participants with abnormal EEG are reported.
Time Frame: EEG taken immediately prior to surgery, during surgery, during cardiovascular intensive care unit (CVICU) stay (up to 48 hours after surgery), and immediately prior to discharge (between 5 to 20 minutes to assess EEG at each time point)
Measure: Count of Participants; unit: Participants
Arm/Group | Narcotic Based Anesthesia | Volatile Anesthesia
Number analyzed (Participants) | 44 | 45
Participants
  Abnormal preoperative EEG | 0 | 0
  Abnormal intraoperative EEG | 1 | 1
  Abnormal EEG in CVICU | 0 | 1
  Abnormal EEG predischarge | 0 | 0

3. Secondary Outcome: Choline
Description: blood levels: time and patient dependent variation, observed patient related trends over time
Time Frame: 0-72 hours
Population: Data were not collected for this outcome measure.
Arm/Group | Narcotic Based Anesthesia | Volatile Anesthesia
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Glutamate
Description: blood levels:time and patient dependent variation, observed patient related trends over time
Time Frame: 0-72 hours
Population: Data were not collected for this outcome measure.
Arm/Group | Narcotic Based Anesthesia | Volatile Anesthesia
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: N-acetylaspartate (Naa)
Description: blood levels:time and patient dependent variation, observed patient related trends over time
Time Frame: 0-72 hours
Population: Data were not collected for this outcome measure.
Arm/Group | Narcotic Based Anesthesia | Volatile Anesthesia
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Lactate
Description: blood levels:time and patient dependent variation, observed patient related trends over time
Time Frame: 0-72 hours
Population: Data were not collected for this outcome measure.
Arm/Group | Narcotic Based Anesthesia | Volatile Anesthesia
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 48 months
Description: Participants with randomization data are included in the analysis.
Arm/Group | Narcotic Based Anesthesia | Volatile Anesthesia
All-Cause Mortality (participants affected / at risk) | 3/44 | 1/45
Serious Adverse Events (participants affected / at risk) | 7/44 | 10/45
Other Adverse Events (participants affected / at risk) | 0/44 | 0/45
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Narcotic Based Anesthesia (N=44) | Volatile Anesthesia (N=45)
Cardiopulmonary arrest (Cardiac disorders) | 0 | 2
Hypotension (Cardiac disorders) | 1 | 2
Arrythmia (Cardiac disorders) | 4 | 3
Bleeding (Vascular disorders) | 2 | 1
Sepsis (Blood and lymphatic system disorders) | 0 | 1
Metabolic acidosis (Metabolism and nutrition disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2012-03-14): https://cdn.clinicaltrials.gov/large-docs/88/NCT03882788/Prot_SAP_000.pdf